CLINICAL TRIAL: NCT01565122
Title: An Observational, Non-interventional, Multi-national Study in Rheumatoid Arthritis (RA) Patients Treated With Tocilizumab
Brief Title: An Observational Study in Rheumatoid Arthritis Patients Treated With RoActemra/Actemra (Tocilizumab)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28207
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multi-center, observational study will evaluate the clinical practice patterns, efficacy and safety of RoActemra/Actemra (tocilizumab) in patients with rheumatoid arthritis. Data will be collected from each eligible patient initiated on RoActemra/Actemra treatment by their treating physician according to approved label for up to 12 months from start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis
* Patients for whom the treating physician has made the decision to commence RoActemra/Actemra treatment. In Group A RoActemra/Actemra has been prescribed within 8 weeks prior to the enrolment visit. In Group B RoActemra/Actemra has been started more than 8 weeks before inclusion in the study, but not before January 2011

Exclusion Criteria:

* RoActemra/Actemra treatment more than 8 weeks prior to inclusion visit for Group A, before January 2011 for Group B
* Previous RoActemra/Actemra treatment in a clinical trial or for compassionate use
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before starting treatment with RoActemra/Actemra
* History of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients initiated on RoActemra/Actemra treatment
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients on RoActemra/Actemra treatment at 6 months | approximately 2.5 years

SECONDARY OUTCOMES:
Rates of dose modifications/interruptions | approximately 2.5 years
Clinical/demographic patient characteristics at initiation of RoActemra/Actemra treatment | approximately 2.5 years
Efficacy: Response according to joint count evaluation by DAS28/EULAR/SDAI/CDAI/ACR | approximately 2.5 years
Efficacy: Monotherapy versus combination therapy | approximately 2.5 years
Safety: Incidence of adverse events | approximately 2.5 years
Quality of life: Patient global assessment of disease activity/VAS-Fatigue/VAS-Pain scales | approximately 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Finland (10):
  - Helsinki
  - Joensuu
  - Jyväskylä
  - Kuopio
  - Lahti
  - Paimio
  - Riihimäki
  - Rovaniemi
  - Tampere
  - Vaasa